CLINICAL TRIAL: NCT02190409
Title: The Effect Of Platelet Rich Fibrin on Implant Stability
Brief Title: An Invivo Study to Compare the Stability of Dental Implants With or Without Platelet Rich Fibrin Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ELİF ONCU (Other)
Collaborators: Baskent University (Other)
Responsible Party: Sponsor-Investigator, ELİF ONCU, Assist.Prof.Dr., Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: D-KA11/06
Record Dates: First submitted 2014-07-08; First posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Dental Implant
Keywords: Dental Implant,
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Test, Control (Experimental): Test: Minimum two tapered implants (Ankylosis, Dentsply Friadent) were placed to each patient. After surgical preparation of implant sockets, PRF that was prepared preoperatively was placed randomly to one of the sockets (PRF+). Acellular plasma portion of PRF was used to wet the implant placed into the PRF-coated socket Control: Other socket was selected as a control group (No Platelet Rich Fibrin used): In the control group no extra intervention used and the conventional procedure was done. Thus the readings of the experimental arm compared with this control.
  Interventions: Device: Dental implant

INTERVENTIONS:
Device: Dental implant — This longitudinal human clinical trial is designed to measure implant stability with the resonance frequency analyzer (Osstell, Integration Diagnostics AB, Sweden) at time of implant placement and up to 4 weeks post placement. delivered. No further follow-up will be done with the resonance frequency approach
  Other Names: The implant in this protocol; 3.5 mm width and 11 mm length) ANKYLOS C/X dental implants were used (Dentsply, Hanau, Germany

SUMMARY:
The purpose of this study was to evaluate the effects of (Platelet Rich Fibrin) PRF application on implant osseointegration in the early phase of healing.

DETAILED DESCRIPTION:
Objectives:Achieving accelerated implant osseointegration could provide immediate or early loading of implants. Platelet-rich fibrin (PRF) is widely used to accelerate soft and hard tissue healing. Activated platelets in PRF release growth factors resulting in cellular proliferation, collagen synthesis and osteoid production. The aim of this study was to compare the stability of dental implants inserted with one-stage surgical protocol with or without PRF application.

Design: Non-randomized, Active Controlled Trial. Material and Methods: Twenty healthy patients (n=10 test group, n= control group) with adequate alveolar bone, having 2 or more adjacent missing teeth, extracted at least 6 months ago were included in this study. Minimum two tapered implants (Ankylosis, DentsplyFriadent) were placed to each patient. After surgical preparation of implant sockets, PRF that was prepared preoperatively was placed randomly to one of the sockets (PRF+). Acellular plasma portion of PRF was used to wet the implant placed into the PRF-coated socket. Resonance frequency measurements were made by Osstell ISQ after placement of implants, at 1 week and one month postoperatively.

Key Words: Dental implant stability, Platelet Rich Fibrin, Resonance frequency analysis

ELIGIBILITY:
Inclusion Criteria:

* The absence of any lesions in the oral cavity, and sufficient residual bone volume to receive two or more adjacent implants of ≥3.5 mm in diameter and 11.0 mm in length, and extracted at least 6 months ago.

Exclusion Criteria:

* Insufficient bone volume
* Parafunctional habits
* Smoking more than 10 cigarettes per day
* Excessive consumption of alcohol
* Localized radiotherapy of the oral cavity
* Antitumor chemotherapy
* Liver, blood, and kidney diseases
* Immunosuppression
* Current corticosteroid or bisphosphonate use
* Pregnancy
* Mucocutaneous diseases involving oral cavity
* Poor oral hygiene

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Implant Stabilitty Quotient (ISQ) evaluation: analysis of the resonance frequency values 4 week period. | Resonance frequency measurements were made by Osstell ISQ after placement of implants, at 1 week and one month postoperatively.
  The stability of the implants were evaluated with the resonance frequency analysis (RFA) method. The measurements were carried out with Osstell ISQ (Implant Stability Quotient) (Osstell, Göteborg, Sweden) by connecting the transducer (smartpeg) to the implant. Two mesio-distal and bucco-lingual measurements were recorded and mean ISQ values were calculated. The resonance frequency measurements were repeated at first and fourth weeks.

SECONDARY OUTCOMES:
Evaluation of osseointegration in different types of bone | Resonance frequency measurements in different bone types were made by Osstell ISQ after placement of implants, at 1 week and one month postoperatively.
  Evaluation early bone healing and compare stability of different bone type (based on the bone quality determined by the insertion torque value)

CONTACTS AND LOCATIONS:
Overall Officials: ELİF ÖNCÜ, 1, Principal Investigator — NECMETTİN ERBAKAN UNIVERSITY
Locations (1):
- NECMETTIN ERBAKAN University Faculty of Dentistry, Department of Periodontology,, Ankara, Turkey (Türkiye)